CLINICAL TRIAL: NCT03137797
Title: Cohort of Patients Naive of Antiretroviral Treatment at Enrollment
Acronym: COPANA
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS CO9 COPANA
Record Dates: First submitted 2016-08-19; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the short, medium and long-term prognosis for newly diagnosed HIV patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the short, medium and long-term prognosis for newly diagnosed HIV patients.

This study aims to precise the impact of HIV infection treatment on morbidity and mortality, the factors related to treatment response, clinical and biological complications, their consequences, especially lipodystrophy and metabolic abnormalities, associated factors especially genetic, aspects linked to aging.

In addition, the study describes the evolution of patients living conditions and behaviors remotely from their screening, particularly related to sexuality, reproduction, and health inequalities and to study the long-term treatment adherence.

One third of the patients were included in the metabolic disorders module. This module includes additional biological and imaging explorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV-1, with a recent diagnosis (<1 year before enrollment)
* Untreated at the time of enrollment,
* Aged 15 or more
* Agreeing to participate in the cohort.

Exclusion Criteria:

* Under protection(saving) of justice

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients infected with HIV-1, with a recent diagnosis (<1 year before enrollment) and untreated at the time of enrollment, aged 15 or more and agreeing to participate in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2004-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Patients prognosis at short, medium and long term | Up to 12 years

SECONDARY OUTCOMES:
Antiretroviral treatment impact | Up to 12 years
  therapeutical adherence, factors related with treatment response
Aging population | up to 12 years
  Study of caracteristics of the population over 50 years old (quality of life or comorbidities... in questionnaire and autoquestionnaire)
Impact of inflammatory markers on antiretroviral treatment | Up to 12 years
  from blood collection: IL-6, sTNF-R1, sTNF-R2, CD14, CRP
Socio-economic conditions (sexuality, education, reproduction, health inequalities) | Up to 12 years
  Completed in annual questionnaire and auto-quesitonnaire by the patient and the physician

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Meyer, Professor, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Meyer, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boufassa F, Goujard C, Viard JP, Carlier R, Lefebvre B, Yeni P, Bouchaud O, Capeau J, Meyer L, Vigouroux C; ANRS COPANA Cohort Study Group. Immune deficiency could be an early risk factor for altered insulin sensitivity in antiretroviral-naive HIV-1-infected patients: the ANRS COPANA cohort. Antivir Ther. 2012;17(1):91-100. doi: 10.3851/IMP1916. PMID 22267473
- [Background] Dray-Spira R, Legeai C, Le Den M, Boue F, Lascoux-Combe C, Simon A, May T, Goujard C, Meyer L; ANRS-COPANA Cohort Study Group. Burden of HIV disease and comorbidities on the chances of maintaining employment in the era of sustained combined antiretoviral therapies use. AIDS. 2012 Jan 14;26(2):207-15. doi: 10.1097/QAD.0b013e32834dcf61. PMID 22008658
- [Background] Rachas A, Warszawski J, Le Chenadec J, Legeai C, Teglas JP, Goujard C, Rouzioux C, Mandelbrot L, Tubiana R, Meyer L. Does pregnancy affect the early response to cART? AIDS. 2013 Jan 28;27(3):357-67. doi: 10.1097/QAD.0b013e32835ac8bc. PMID 23079802
- [Background] Krastinova E, Seng R, Yeni P, Viard JP, Vittecoq D, Lascoux-Combe C, Fourn E, Pahlavan G, Delfraissy JF, Goujard C, Meyer L; ANRS PRIMO and COPANA Cohorts. Is clinical practice concordant with the changes in guidelines for antiretroviral therapy initiation during primary and chronic HIV-1 infection? The ANRS PRIMO and COPANA cohorts. PLoS One. 2013 Aug 1;8(8):e71473. doi: 10.1371/journal.pone.0071473. Print 2013. PMID 23936509
- [Background] Legeai C, Vigouroux C, Souberbielle JC, Bouchaud O, Boufassa F, Bastard JP, Carlier R, Capeau J, Goujard C, Meyer L, Viard JP; ANRS-COPANA Cohort Study Group. Associations between 25-hydroxyvitamin D and immunologic, metabolic, inflammatory markers in treatment-naive HIV-infected persons: the ANRS CO9 <<COPANA>> cohort study. PLoS One. 2013 Sep 18;8(9):e74868. doi: 10.1371/journal.pone.0074868. eCollection 2013. PMID 24058636
- [Background] Boufassa F, Lechenadec J, Meyer L, Costagliola D, Hunt PW, Pereyra F, Deeks S, Pancino G, Taulera O, Lichterfeld M, Delobel P, Saez-Cirion A, Lambotte O; ANRS CO18 HIV Controllers Cohort; Cascade Collaboration in Eurocoord; SCOPE Cohort; International HIV Controllers Study. Blunted response to combination antiretroviral therapy in HIV elite controllers: an international HIV controller collaboration. PLoS One. 2014 Jan 17;9(1):e85516. doi: 10.1371/journal.pone.0085516. eCollection 2014. PMID 24465584
- [Background] El Khoury P, Ghislain M, Villard EF, Le Goff W, Lascoux-Combe C, Yeni P, Meyer L, Vigouroux C, Goujard C, Guerin M. Plasma cholesterol efflux capacity from human THP-1 macrophages is reduced in HIV-infected patients: impact of HAART. J Lipid Res. 2015 Mar;56(3):692-702. doi: 10.1194/jlr.M054510. Epub 2015 Jan 8. PMID 25573889
- [Background] Ghislain M, Bastard JP, Meyer L, Capeau J, Fellahi S, Gerard L, May T, Simon A, Vigouroux C, Goujard C; ANRS-COPANA Cohort Study Group. Late Antiretroviral Therapy (ART) Initiation Is Associated with Long-Term Persistence of Systemic Inflammation and Metabolic Abnormalities. PLoS One. 2015 Dec 4;10(12):e0144317. doi: 10.1371/journal.pone.0144317. eCollection 2015. PMID 26636578
- [Background] Ploquin MJ, Madec Y, Casrouge A, Huot N, Passaes C, Lecuroux C, Essat A, Boufassa F, Jacquelin B, Jochems SP, Petitjean G, Angin M, Gartner K, Garcia-Tellez T, Noel N, Booiman T, Boeser-Nunnink BD, Roques P, Saez-Cirion A, Vaslin B, Dereudre-Bosquet N, Barre-Sinoussi F, Ghislain M, Rouzioux C, Lambotte O, Albert ML, Goujard C, Kootstra N, Meyer L, Muller-Trutwin MC. Elevated Basal Pre-infection CXCL10 in Plasma and in the Small Intestine after Infection Are Associated with More Rapid HIV/SIV Disease Onset. PLoS Pathog. 2016 Aug 10;12(8):e1005774. doi: 10.1371/journal.ppat.1005774. eCollection 2016 Aug. PMID 27509048